CLINICAL TRIAL: NCT02806479
Title: Pilot Observational Case-control Study of the Electrical Heterogeneity in Patients With Hypertrophic Cardiomyopathy and High Arrhythmic Risk
Brief Title: Hypertrophic Cardiomyopathy Pilot Study
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Larisa Tereshchenko, Assistant Professor, Oregon Health and Science University
Other Study IDs: 15049
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hypertrophic Cardiomyopathy; Coronary Artery Disease
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Case: Hypertrophic cardiomyopathy: HCM patients at high risk for ventricular arrhythmia
  Interventions: Other: Observational: Arrhythmogenic Substrate
- Control I: Healthy: Healthy Controls
- Control II: Post-MI with arrhythmogenic substrate: Ischemic cardiomyopathy patients with documented history of ventricular tachyarrhythmia and left ventricular hypertrophy
  Interventions: Other: Observational: Arrhythmogenic Substrate
- Control III: VT/VF-free ischemic cardiomyopathy: Ischemic cardiomyopathy patients without ventricular arrhythmia, as proven by non-inducibility and history of freedom from ventricular tachyarrhythmia during at least one ICD generator life

INTERVENTIONS:
Other: Observational: Arrhythmogenic Substrate
  Groups: Case: Hypertrophic cardiomyopathy; Control II: Post-MI with arrhythmogenic substrate

SUMMARY:
This study evaluates mechanisms of arrhythmogenicity in hypertrophic cardiomyopathy, in comparison to patients with well-understood arrhythmogenic substrate (ischemic cardiomyopathy), as well as to individuals free from arrhythmogenic substrate

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HCM
* Documented history of sustained ventricular tachyarrhythmia or resuscitated sudden cardiac arrest
* Maximal left ventricular wall thickness of > 30mm
* Extensive fibrosis on cardiac MRI (>15% of total myocardial volume)
* >7.5%/5-year risk of sudden cardiac death as determined by HCM risk-SCD

Exclusion Criteria:

* age < 18 years
* Pregnancy
* Atrial Fibrillation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case - Control study of hypertrophic cardiomyopathy patients at high risk for ventricular arrhythmias in comparison to three Controls groups
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Non-invasively reconstructed epicardial activation map | within one day

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perez-Alday EA, Haq KT, German DM, Hamilton C, Johnson K, Phan F, Rogovoy NM, Yang K, Wirth A, Thomas JA, Dalouk K, Fuss C, Ferencik M, Heitner S, Tereshchenko LG. Mechanisms of Arrhythmogenicity in Hypertrophic Cardiomyopathy: Insight From Non-invasive Electrocardiographic Imaging. Front Physiol. 2020 Apr 24;11:344. doi: 10.3389/fphys.2020.00344. eCollection 2020. PMID 32390862